CLINICAL TRIAL: NCT06546137
Title: National Network for Cardiovascular Genomics: Advancing Cardiovascular Healthcare for Hereditary Diseases in Brazil's Unified Health System Through a Multicenter Registry
Acronym: RENOMICA-Hcor
Status: Recruiting | Type: Observational
Sponsor: Hospital do Coracao (Other)
Collaborators: Instituto Nacional de Cardiologia de Laranjeiras (Other); Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Sponsor
Other Study IDs: RENOMICA-Hcor
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-11

CONDITIONS: Cardiomyopathy, Hypertrophic; Cardiomyopathy, Dilated; Cardiomyopathy Restrictive; Arrhythmogenic Right Ventricular Dysplasia; Non-Compaction Cardiomyopathy; Familial Hypercholesterolemia; Marfan Syndrome; Ehlers-Danlos Syndrome, Vascular Type; Loeys-Dietz Syndrome; Long QT Syndrome; Short Qt Syndrome; Brugada Syndrome; Catecholaminergic Polymorphic Ventricular Tachycardia; Sudden Cardiac Death
Keywords: hereditary cardiovascular diseases; whole genome sequencing
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Cardiomyopathy, Dilated; Cardiomyopathy, Restrictive; Arrhythmogenic Right Ventricular Dysplasia; Hyperlipoproteinemia Type II; Marfan Syndrome; Ehlers-Danlos Syndrome, Type IV; Loeys-Dietz Syndrome; Long QT Syndrome; Short Qt Syndrome; Brugada Syndrome; Polymorphic Catecholaminergic Ventricular Tachycardia; Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Saliva or cheek swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: whole genome sequencing — whole genome sequencing of genomic DNA extracted from buccal swab

SUMMARY:
The goal of this observational study is to develop a registry of Brazilian patients with hereditary cardiovascular diseases, combining clinical and genomic data. The main questions it aims to answer are:

Which genes are most commonly affected? What is the frequency of these genetic alterations in our population? Participants will be interviewed in routine medical care visits and their DNA will be sequenced.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of a hereditary cardiovascular disease according to current clinical guidelines
* Agree to receive genetic counseling
* Sign informed consent form
* Provide the information required in the case report form

Exclusion Criteria:

* Signature absent from informed consent form
* Inadequate buccal swab (sample may be collected twice)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients under routine medical care in hospitals and clinics located in Brazil with a clinical diagnosis of an hereditary cardiovascular disease.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield | 30 months after study start date
  Percentage of participants with pathogenic or likely pathogenic variants
Genetic diversity | 30 months after study start date
  Determine genes that cause hereditary cardiovascular diseases in Brazil
Variant frequency | 30 months after study start date
  Determine the frequency of disease-causing and benign variants in the Brazilian population

CONTACTS AND LOCATIONS:
Locations (27):
- Brazil (27):
  - Centro de Pesquisa Silvestre Santé, Rio Branco, Acre
  - Centro de Pesquisas Clínicas Dr. Marco Mota, Maceió, Alagoas
  - Hospital Universitário da Unifap, Macapá, Amapá
  - Hospital de Messejana Dr. Carlos Alberto Studart Gomes, Fortaleza, Ceará
  - Hospital Universitário Professor Edgard Santos, Salvador, Estado de Bahia
  - Hospital Ana Nery - HAN/SESAB, Salvador, Estado de Bahia
  - Instituto de Cardiologia e Transplantes do Distrito Federal, Brasília, Federal District
  - Hospital das Clínicas da Universidade Federal de Goiás - HC-UFG, Goiânia, Goiás
  - Universidade Ceuma, São Luís, Maranhão
  - Hospital Felicio Rocho - HFR, Belo Horizonte, Minas Gerais
  - Liga Mineira de Ressuscitação Cardiopulmonar, Belo Horizonte, Minas Gerais
  - Santa Casa de Misericórdia de Montes Claros, Montes Claros, Minas Gerais
  - Health & Care, Belém, Pará
  - Hospital Universitário Pedro Ernesto - UERJ, Rio de Janeiro, Rio de Janeiro
  - Instituto de Puericultura e Pediatria Martagão Gesteira, Rio de Janeiro, Rio de Janeiro
  - Hospital Universitário Clementino Fraga Filho - UFRJ, Rio de Janeiro, Rio de Janeiro
  - Instituto Nacional de Cardiologia, Rio de Janeiro, Rio de Janeiro
  - Hospital Universitário Onofre Lopes - UFRN, Natal, Rio Grande do Norte
  - Hospital das Clínicas de Porto Alegre - UFRGS, Porto Alegre, Rio Grande do Sul
  - Instituto de Cardiologia - Fundação Universitária de Cardiologia de Porto Alegre - IC-FUC, Porto Alegre, Rio Grande do Sul
  - Instituto de Pesquisa e Ensino em Saúde - IPES, Porto Velho, Rondônia
  - Hospital Universitário Professor Polydoro Ernani de São Thiago - UFSC, Florianópolis, Santa Catarina
  - Centro Multidisciplinar de Ensino Especializado e Pesquisa Ltda, Joinville, Santa Catarina
  - Hospital Universitário São Francisco na Providência de Deus, USF-SP, Bragança Paulista, São Paulo
  - Hospital Universitário da Universidade Federal de São Carlos, São Carlos, São Paulo
  - Hospital do Coracao, São Paulo, São Paulo
  - Universidade Federal do Tocantins, Palmas, Tocantins

IPD SHARING:
Plan to Share IPD: No
Genomic data are sensitve and will not be shared for individual participants